CLINICAL TRIAL: NCT03734068
Title: Observational Prospective Study on Chemoembolization Using LifePearl Polyethylene Glycol Drug Eluting Microspheres With Doxorubicin in Patients With Primary Un-resectable Liver Cancer (Hepatocellular Carcinoma)
Brief Title: Chemoembolization Using LifePearl Polyethylene Glycol Drug Eluting Microspheres With Doxorubicin in HCC
Acronym: LIFDOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Group of Endovascular Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: LIFDOX
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Tumor response; Lifepearls
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemoembolization: Chemoembolization Using LifePearl and Doxorubicin
  Interventions: Device: Chemoembolization Using LifePearl; Drug: Doxorubicin

INTERVENTIONS:
Device: Chemoembolization Using LifePearl — Chemoembolization Using LifePearl
Drug: Doxorubicin — Doxorubicin is loaded to LIfePearl

SUMMARY:
The aim of this study is to collect data on efficacy and tolerability on a large series of patient of different Italian hospitals in order to support the validation of LifePearl with robust and consistent clinical evidence. Since TACE in treating HCC is considered a more common and accepted approach, this study will be focused on evaluating treatment efficacy and safety of LIFDOX for un-resectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common type of cancer in men and the seventh in women and is the third most common cause of death from cancer worldwide. The overall incidence of HCC remains high in developing countries and is steadily increasing in most industrialized countries.

Trans-arterial chemoembolization (TACE) is the most used treatment for patients with un-resectable hepatocellular carcinoma (HCC), because it improves median survival and tumor response. The application of drug-eluting bead to this procedure has significantly increased TACE efficacy, while reducing systemic drug leakage, liver toxicity and adverse events. These beads deliver the toxic drugs directly to the arterial capillary bed of the tumor, and release them in a controlled manner. This method lower the systemic exposure to chemotherapeutics, while increasing their local concentration, resulting in a greater tissue necrosis than classic trans-arterial chemoembolization.

TACE is indicated for patients with multinodular liver cancer that have no vascular invasion and extrahepatic diffusion. TACE is also strongly suggested for patients with un-resectable liver primary tumor (HCC and cholangiocarcinoma) and chemo-resistant liver metastases, mainly from colorectal cancer carcinoma (CRC), and is widely performed in 32% of patients with un-resectable HCC at initial diagnosis and in 58% of those with recurrent HCC. It appears, moreover, to be particularly useful if carried out with new embolization materials, such as doxorubicin.

Trans-arterial chemoembolization is constantly improving; from the original conventional TACE using Lipiodol and sponge particles, some years ago it evolved into precision TACE, thanks to the availability of drug-eluting microspheres. Microspheres retain the ability to bind positively charged chemotherapeutic drugs (i.e.: doxorubicin) and release them in a prolonged and sustained kinetic at tumor site while determining a permanent embolization of the feeding arteries. Consequently, less systemic exposure of drug is observed, with a benefit for the patients in term of toxicity, quality of life and hospitalization.

Recently, new drug-eluting beads in polyethylene glycol has been made available, termed LifePearl Polyethylene glycol drug eluting microspheres (Terumo, Microvention, Tustin, CA, USA), which are offered as a syringe presentation, for an easier loading process. More interestingly, LifePearl are precisely calibrated, in a range ≤ 50 micron, potentially leading to a more distal and targeted distribution into the tissues; in addition, they are endowed with a prolonged time in suspension after dilution in contrast medium, which makes the administration more smooth, predictable and reproducible. Because of the above improvements, LifePearl are now widely used in several hospital for the Transarterial chemoembolization as everyday clinical practice, for the hepatic intra-arterial infusion of doxorubicin or irinotecan respectively for the therapy of primary and metastatic liver cancer.

The aim of this study is to collect data on efficacy and tolerability on a large series of patient of different Italian hospitals in order to support the validation of LifePearl with robust and consistent clinical evidence. Since TACE in treating HCC is considered a more common and accepted approach, this study will be focused on evaluating treatment efficacy and safety of LIFDOX for un-resectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of HCC with CT scan, MRI or biopsy
* Patient with un-resectable HCC and not indicated for other radical therapies, or waiting for transplant
* Multinodular or single nodular tumor extended to <50% of the liver
* Hyper vascular lesion showing contrast enhancement in the early stage at the contrast media bolus injection CT or MRI.
* At least one uni-dimensional lesion measurable according to the Modified RECIST criteria by CT-scan or MRI
* No invasion in the blood vessel (hepatic portal, hepatic vein) or bile duct by the CT or MR
* Eastern Cooperative Oncology Group performance status is 0 - 1
* Proper blood, liver, renal, heart function
* Over 18 years old
* Expected survival more than 6 months
* Prior written patient consent

Exclusion Criteria:

* Extrahepatic metastasis (Any lymph nodes measuring ≥ 10mm along the short axis)
* Tumor burden involving more than 50% of the liver
* History of biliary tract repair or endoscopic biliary tract treatment
* Clinically important refractory ascites or pleural fluid
* Any contraindications for hepatic embolization procedures
* Any contraindication for doxorubicin administration
* Contrast media allergy contraindicating angiography
* Acute or active cardiac, hepatic or renal diseases
* Pregnant, nursing or childbearing age women and men who are sexually active and don't want to or can't do contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: un-resectable hepatocellular carcinoma that are indicated for TACE treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 6 months
  CT scan will be performed to assess tumor response

SECONDARY OUTCOMES:
Number of adverse events | 1 year
  number and intensity of adverse events will be monitored
time to progression | 1 months
  time from first treatment to progression will be computed
number of treatment required to achieve objective response in HCC patients | 1 year
  number of treatment required to achieve objective response (partial or complete response) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Nicolini, MD, Principal Investigator — UOSD Radiologia Interventistica, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Via Francesco Sforza, 28, 20122 Milano, Italia; Giammaria Fiorentini, MD, Study Chair — Department of Oncology-Hematology, Azienda Ospedaliera Ospedali Riuniti Marche Nord, P.O. San Salvatore, via C. Lombroso 1, 62122 Pesaro, Italy
Locations (1):
- Antonio Nicolini, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The researchers will provide full protocol to interested researchers
Supporting Information: Study Protocol
Time Frame: 12 months
Access Criteria: request by email to Principal investigator